CLINICAL TRIAL: NCT03371836
Title: Use of Clobazam in Treating Anxiety Comorbid With Pediatric Epilepsy
Brief Title: Use of Clobazam for Epilepsy and Anxiety
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Principal Investigator, Jay Salpekar, M.D., Principal Investigator, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: onfi90037
Record Dates: First submitted 2017-11-21; First posted 2017-12-13 (Actual); Results first posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Epilepsy; Anxiety
Keywords: pediatrics
MeSH Terms: conditions — Epilepsy; Anxiety Disorders | interventions — Clobazam

STUDY DESIGN:
Intervention Model Description: All participants receive treatment and outcome is assessed; there is no control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Clobazam (Other): open label (single treatment arm)
  Interventions: Drug: Clobazam

INTERVENTIONS:
Drug: Clobazam — Clobazam is used as an adjunct medicine for all participants.
  Other Names: Onfi

SUMMARY:
This study is an open label, adjunctive, proof of concept, pilot clinical trial. Pediatric patients with epilepsy and clinically significant anxiety will be recruited and if enrolled will receive active treatment, involving flexible dose titration of clobazam and will be monitored for a period of four months. The study will be monitored and overseen by the Johns Hopkins Hospital Institutional Review Board.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of epilepsy, characterized by focal seizures with suspected or documented localization in the temporal lobe. All participants will have active epilepsy that requires treatment with anticonvulsant medication.

  * Although it is not necessary to be seizure free, a seizure baseline period will be established in the 60 days prior to enrollment into the study.
  * Current regimen of anticonvulsant drugs must have been stable for 30 days prior to entry into the study.
* No episodes of seizure clusters of status epilepticus within 30 days prior to entry into the study.
* Established symptoms of anxiety with functional impairment.
* A diagnosis of an anxiety disorder based on the administration of the K-SADS Male or female participants equal to or above age 6 and below age 18 at the start of the study. No exclusion will be made on the basis of gender or minority status.
* Male or female participants equal to or above age 6 and below age 18 at the start of the study. No exclusion will be made on the basis of gender or minority status.
* Good general health as determined by medical history and physical examination.
* Ability to swallow pills (participant will receive pill swallowing instruction if necessary). The medicine may be cut into pieces and/or mixed with applesauce.
* If female of childbearing age, a negative urine or serum pregnancy test must be established or assured at baseline. Additionally, the participant must agree to use abstinence or appropriate contraception methods or be otherwise incapable of pregnancy for the duration of the study. Pregnancy test results will be shared with parent or guardian. Pregnancy status (or prevention) and abstinence or contraception methods will be addressed throughout the study for females of childbearing age as well as for post-pubertal males.
* Previous subjects who failed at any point to meet continuation criteria and withdrew early may be considered for re-enrollment by the PI on a case-by-case basis.
* Participant or legal caregiver capable of providing informed consent and fully capable of monitoring the subject's disease process and compliance with treatment.

Exclusion criteria:

* Previous allergic or hypersensitivity reactions to Onfi® or benzodiazepines
* Active substance abuse or dependence within 30 days of enrollment
* DSM-V diagnosis of psychotic illness or imminent risk of harm to self or others.
* Current standing use of benzodiazepines (except as "rescue" medicine)
* Serious or unstable medical or neurologic conditions such as HIV, liver or kidney disease, cancer or diabetes.
* Participation in a previous experimental drug study within 30 days of baseline visit.
* Estimated IQ<70 as indicated by initial clinical assessment (rendering rating scales invalid)
* Insufficient capacity of caregiver or legal guardian to understand and appropriately consent for study procedures

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Salpekar, MD, Principal Investigator — KKI/JH
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Clobazam: open label single treatment arm
  Clobazam is used as an adjunct medicine for all participants.
Period: Overall Study
Arm/Group | Clobazam
Started | 20
Completed | 18
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Open Label Single Treatment Arm: open label
  Clobazam: Clobazam is used as an adjunct medicine for all participants.
Arm/Group | Open Label Single Treatment Arm
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 13.8 [6 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: CGI-I
Description: Mean of Clinical Global Impression-Improvement from baseline. (1-7 point scale; lower score equals a better outcome; 1 is the maximum improvement, 7 is the minimum improvement)
Time Frame: 14-18 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Clobazam
Number analyzed (Participants) | 18
units on a scale | 2 [1 to 7]

ADVERSE EVENTS:
Time Frame: up to 18 weeks
Arm/Group | Open Label Single Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT03371836/Prot_SAP_000.pdf